CLINICAL TRIAL: NCT04696809
Title: A Phase 1/2 Study of JNJ-64007957, a Humanized BCMA * CD3 Bispecific Antibody in Japanese Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Teclistamab in Japanese Participants With Relapsed or Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108949; 64007957MMY1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-01-05; First posted 2021-01-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Japanese Participants with Relapsed or Refractory Multiple Myeloma (MM) (Experimental): Japanese participants will receive Teclistamab subcutaneously (SC) at four dose levels. Cohort 1 will receive Teclistamab at Dose 1 and 2 (step-up doses) prior to first treatment dose on Day 1 followed by Dose 3 weekly (that is, on Days 1,8, and 15 of a 21-day cycle). Cohort 2 will receive Teclistamab at Dose 1 and 4 (step up doses) prior to first treatment dose on Day 1 followed by Dose 5 weekly. Cohort 3 will receive Teclistamab at Dose 1, 4, and 5 (step up doses) prior to first treatment dose on Day 1 followed by Dose 6 weekly. Cohort 4 will receive Teclistamab at Dose 1, 4, and 5 (step up doses) prior to first treatment dose on Day 1 followed by Dose 7 weekly for (2 cycles), then biweekly (cycle 3 to 6) on Days 1 and 15 and monthly (cycle 7) on Day 1 of 1 28-day cycle. In Phase 2 , participants will receive Teclistamab SC at Dose 1 and 4 (step up doses) up to 8 days prior to first treatment dose on Day 1 followed by Dose 5 on Days 1,8,15, and 22 of a 28-day cycle.
  Interventions: Drug: Teclistamab

INTERVENTIONS:
Drug: Teclistamab — Teclistamab will be administered subcutaneously.
  Other Names: JNJ-64007957

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability in Japanese participants with relapsed or refractory multiple myeloma (RRMM) at the recommended Phase 2 dose (RP2D) identified in Study 64007957MMY1001 (NCT03145181) in Phase 1 part and to evaluate the efficacy of teclistamab at RP2D for Japanese participants in Phase 2 part.

ELIGIBILITY:
Inclusion criteria:

* Documented diagnosis of multiple myeloma (MM) according to International Myeloma Working Group (IMWG) diagnostic criteria
* Participant must have measurable disease defined by any of the following: Serum M-protein level greater than or equal to (>=) 1.0 gram per deciliter (g/dL); Urine M-protein level >= 200 milligrams per 24 hours (mg/24 hours); or Light chain MM, for participants without measurable disease in the serum or urine: serum Ig-free light chain (FLC) >=10 milligrams per deciliter (mg/dL) and abnormal serum Ig kappa-lambda FLC ratio; or if central laboratory assessments are not available, relevant local laboratory measurements must exceed the minimum required level by at least 25 percent (%)
* Participant must be relapsed or refractory to established therapies with known clinical benefit in relapsed/refractory MM or be intolerant to established MM therapies and a candidate for teclistamab treatment in the opinion of the treating physician. Prior lines of therapy must include a proteasome inhibitors (PI), an immunomodulatory drug (IMiD), and an anti-CD38 antibody in any order during the course of treatment. Participants who could not tolerate PI, immunomodulatory drugs, or anti-CD38 antibody are allowed
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1 at screening and immediately before the start of study treatment administration
* Woman of childbearing potential must have a negative pregnancy test at screening and within 24 hours prior to the first dose of study treatment using highly sensitive pregnancy test either serum (beta-human chorionic gonadotropin [beta-hCG]) or urine

Exclusion criteria:

* Prior treatment with any B cell maturation antigen (BCMA)-targeted therapy
* Toxicities from previous anticancer therapies that have not resolved to baseline levels or to less than or equal to (<=) Grade 1 except for alopecia or peripheral neuropathy
* Received a cumulative dose of corticosteroids equivalent to >=140 mg of prednisone within the 14-day period before the first step-up dose of study treatment (does not include pretreatment medication)
* Stem cell transplantation: An allogeneic stem cell transplant within 6 months. Participants who received an allogeneic transplant must be off all immunosuppressive medications for 6 weeks without signs of graft-versus-host disease; Received an autologous stem cell transplant less than or equal (<=) 12 weeks before the first step-up dose of study treatment
* Central nervous system involvement or clinical signs of meningeal involvement of MM. If either is suspected, whole brain magnetic resonance imaging (MRI) and lumbar cytology are required during screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2026-04-22 (Estimated); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of Participants with Adverse Events (AE) | Up to 1 year and 5 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non investigational) product.
Phase 1: Number of Participants with Serious Adverse Events (SAE) | Up to 1 year and 5 months
  A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Phase 1: Number of Participants with Dose Limiting Toxicity (DLT) | Up to 28 days
  Number of participants with DLT will be assessed. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.
Phase 2: Overall response rate (ORR) | Up to 1 year and 5 months
  ORR is defined as the percentage of participants who have a partial response (PR) or better according to the 2016 International Myeloma Working Group (IMWG) response criteria.

SECONDARY OUTCOMES:
Phase 1 and Phase 2: Serum Concentration of Teclistamab | Up to 1 year and 5 months
  Serum concentration of Teclistamab will be assessed.
Phase 1: Systemic Cytokine Concentrations | Up to 1 year and 5 months
  Cytokines concentration will be measured for biomarker assessment.
Phase 1 and Phase 2: Number of Participants with Anti-teclistamab Antibodies | Up to 1 year and 5 months
  Number of participants with anti-teclistamab antibodies will be assessed.
Phase 1: Objective Response Rate | Up to 1 year and 5 months
  Objective response will be defined as partial response (PR) or better as defined by the 2016 IMWG response criteria in multiple myeloma (MM).
Phase 1 and Phase 2: Duration of Response (DOR) | Up to 1 year and 5 months
  DOR is defined as the duration from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the 2016 IMWG criteria, or death.
Phase 1 and Phase 2: Time to Response (TTR) | Up to 1 year and 5 months
  TTR is defined as the time between date of first dose of study treatment and the first efficacy evaluation that the participant has met all criteria for PR or better.
Phase 2: Very Good Partial Response (VGPR) or Better Response Rate (Stringent Complete Response [sCR]+ Complete Response [CR]+VGPR) | Up to 1 year and 5 months
  VGPR or better response rate (sCR+CR+VGPR) is defined as the percentage of participants who achieve a VGPR or better response according to the 2016 IMWG response criteria.
Phase 2: Complete Response (CR) or Better Response Rate | Up to 1 year and 5 months
  CR or better response rate is defined as the percentage of participants who achieve a CR or better response (sCR+CR) according to the IMWG 2016 criteria.
Phase 2: Stringent Complete Response (sCR) Rate | Up to 1 year and 5 months
  sCR rate is defined as the percentage of participants who achieve an sCR according to the IMWG 2016 criteria.
Phase 2: Progression-free Survival (PFS) | Up to 1 year and 5 months
  PFS is defined as the time from the date of first dose of study drug to the date of first documented disease progression, as defined in the 2016 IMWG response criteria, or death due to any cause, whichever occurs first.
Phase 2: Overall survival (OS) | Up to 1 year and 5 months
  OS is defined as the time from the date of first dose of study drug to the date of the participant's death. If the participant is alive or the vital status is unknown, then the participant's data will be censored at the date the participant was last known to be alive.
Phase 2: Minimal Residual Disease (MRD)-negative Rate | Up to 1 year and 5 months
  MRD-negative rate is defined as the percentage of participants who achieved MRD-negative status to a threshold of 10^-5 at any timepoint after initial dose of teclistamab and before disease progression or starting subsequent therapy.
Phase 2: Number of Participants with AEs | Up to 1 year and 5 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non investigational) product.
Phase 2: Number of Participants with AEs by Severity | Up to 1 year and 5 months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 with the exception of cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS), which will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) guidelines. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Phase 2: Number of Participants with SAEs | Up to 1 year and 5 months
  A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Phase 2: Number of Participants with SAEs by Severity | Up to 1 year and 5 months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 with the exception of cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS), which will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) guidelines. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Phase 2: Number of Participants with Abnormalities in Clinical Laboratory Test Values | Up to 1 year and 5 months
  Number of participants with abnormalities in clinical laboratory test values of hematology, serum chemistry, and coagulation will be reported.
Phase 2: Number of Participants with Abnormalities in Clinical Laboratory Test Values by Severity | Up to 1 year and 5 months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 with the exception of cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS), which will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) guidelines. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Phase 2: Change from Baseline in Health-related Quality of Life (HRQoL) (Symptoms, Functioning, and Well-being) Assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30) Score | Up to 1 year and 5 months
  Change from baseline in EORTC- QLQ-C30 score will be reported. The EORTC- QLQ-C30 Version 3 includes 30 items that make up 5 functional scales (physical, role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (pain, fatigue, and nausea/vomiting), and 6 single symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The item and scale scores are transformed to a 0 to 100 scale. A higher score represents greater HRQoL, better functioning, and more (worse) symptoms.
Phase 2: Change from Baseline in EuroQol Five Dimension Five Level Questionnaire (EQ-5D-5L) Scale | Up to 1 year and 5 months
  Change from baseline in EQ-5D-5L scale will be reported. The EQ-5D-5L is a generic measure of health status. EQ-5D-5L is a 5 item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Phase 2: Change from Baseline in Patient Global Impression of Severity (PGIS) Scale | Up to 1 year and 5 months
  Change from baseline in PGIS scale will be reported. The PGIS is a single item that assesses severity of the participant's health state, on a 5-point verbal rating scale (1: None, 2: Mild, 3: Moderate, 4: Severe, 5: Very Severe) at the time of completing the PRO measure. Higher score indicate greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical trials, Study Director — Janssen Pharmaceutical K.K.
Locations (15):
- Japan (15):
  - Kameda Medical Center, Chiba
  - Ogaki Municipal Hospital, Gifu
  - National Hospital Organization Mito Medical Center, Higashiibaraki-gun
  - Kobe City Medical Center General Hospital, Kobe
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Kurume University Hospital, Kurume
  - Kyoto Kuramaguchi Medical Center, Kyoto
  - National Hospital Organization Matsumoto Medical Center, Matsumoto
  - Nagoya City University Hospital, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - National Hospital Organization Okayama Medical Center, Okayama
  - Osaka International Cancer Institute, Osaka
  - Japanese Red Cross Osaka Hospital, Osaka
  - National Hospital Organization Hiroshima-Nishi Medical Center, Ōtake
  - Japanese Red Cross Medical Center, Shibuya City

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Martin TG, Mateos MV, Yi JH, van de Donk NWCJ, Cai Z, Fu W, Garfall AL, Iida S, Jung SH, Kuroda Y, Niu T, Nooka AK, Min CK, Sidana S, Chastain K, Doyle M, Nishikawa K, Wang X, Song Y, Yamazaki H, Izumi Y, Zhuo J, Zhu A, Yoon DH, Du J, Ishida T. Efficacy and safety of teclistamab in triple-class exposed relapsed/refractory multiple myeloma: Pooled findings from three clinical cohorts and a retrospective cohort. Cancer. 2026 Jan 1;132(1):e70237. doi: 10.1002/cncr.70237. PMID 41485109